CLINICAL TRIAL: NCT05053386
Title: A Randomized Controlled, Multi-center Clinical Study of Anbijian (Idarubicin Hydrochloride for Injection) vs. Epirubicin Lipiodol Emulsion Transhepatic Arterial Chemoembolization in the Treatment of Hepatocellular Carcinoma
Brief Title: Idarubicin vs. Epirubicin TACE in the Treatment of Hepatocellular Carcinoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, guoliang shao, A Randomized Controlled, Multi-center Clinical Study of Anbijian (Idarubicin Hydrochloride for Injection) vs. Epirubicin Lipiodol Emulsion Transhepatic Arterial Chemoembolization in the Treatment of Hepatocellular Carcinoma, Zhejiang Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-2021-208
Record Dates: First submitted 2021-09-13; First posted 2021-09-22 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Idarubicin; Injections; Epirubicin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Idarubicin (Experimental): 10mg idarubicin is dissolved in 5ml water for injection, and 5~20ml lipiodol is used to prepare lipiodol emulsion.
  Interventions: Drug: Idarubicin Hydrochloride for Injection
- Epirubicin (Active Comparator): 50mg epirubicin is dissolved in 5ml 5% glucose solution, and 5~20ml lipiodol is used to prepare lipiodol emulsion.
  Interventions: Drug: Epirubicin

INTERVENTIONS:
Drug: Idarubicin Hydrochloride for Injection — After an interventional treatment, CT and/or MRI, tumor-related markers, liver and kidney function and blood routine examinations will be reviewed every 4-6 weeks, based on the patient's response to the last treatment, changes in liver function and physical fitness, and CT And (or) dynamic enhanced MRI scan to evaluate the survival of liver tumors and determine the next TACE treatment. At least 2 cycles are applied and no more than 4 cycles are applied.
  Other Names: Anbijian
  Arms: Idarubicin
Drug: Epirubicin — After an interventional treatment, CT and/or MRI, tumor-related markers, liver and kidney function and blood routine examinations will be reviewed every 4-6 weeks, based on the patient's response to the last treatment, changes in liver function and physical fitness, and CT And (or) dynamic enhanced MRI scan to evaluate the survival of liver tumors and determine the next TACE treatment. At least 2 cycles are applied and no more than 4 cycles are applied.
  Other Names: Epirubicin Hydrochloride
  Arms: Epirubicin

SUMMARY:
In this study, patients with hepatocellular carcinoma were used as the research object to explore the effectiveness and safety of idarubicin hepatic artery perfusion combined with lipiodol embolization, and to preliminarily explore the possibility of idarubicin in the treatment of hepatocellular carcinoma. Provide evidence-based medicine for the discovery of better TACE combined chemotherapy regimens for the treatment of hepatocellular carcinoma.

DETAILED DESCRIPTION:
China is a country with a high incidence of liver cancer, the annual incidence of nearly 50% of the world. At present, transcatheter Arterial chemoembolization (TACE) has become one of the main treatment methods for primary liver cancer and liver metastasis, and has been recognized as the first choice for inoperable primary liver cancer. In addition, it has also been applied in the treatment of resectable liver cancer, liver cancer with tumor embolus and liver metastasis, which is safe and reliable.

Idarubicin is a DNA topoisomerase II inhibitor that promotes DNA strand breakage, trapping cells in the G2 phase of the cell cycle, DNA cleavage, and cell apoptosis. At the same time, it can be inserted between the DNA base pairs and create freedom. Preclinical studies have shown that Idarubicin has superior antitumor activity than epirubicin, especially against SUN-449 human hepatoma cells. In recent years, foreign scholars have conducted a series of explorations in the treatment of hepatocellular carcinoma with Idarubicin TACE, and have obtained positive results.

This study aims to evaluate the safety and effectiveness of idarubicin lipiodol emulsion hepatic artery chemoembolization in the treatment of hepatocellular carcinoma, in order to provide evidence-based medical evidence for the discovery of a better TACE treatment regimen for advanced hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

18-80 years old, no gender limit; Confirmed as hepatocellular carcinoma by histopathology or clinical diagnosis; The expected survival period is ≥3 months; Chinese liver cancer staging program (CNLC) IIb/IIIa, liver function Child pugh A or B, or Surgical resection, but due to other reasons (such as advanced age, severe liver cirrhosis, etc.) unable or unwilling to receive surgical treatment CNLC stage Ib and IIa liver cancer patients; ECOG score 0-1 points; At least one measurable lesion (spiral CT scan ≥10mm); Laboratory inspection indicators meet the following requirements: Peripheral blood: WBC≥4.0×109/L，PLT≥80×109/L，Hb≥90g/L. Renal function: Cr≤2.0×UNL (upper limit of normal); Liver function: BIL≤2.0×UNL (upper limit of normal), ALT/AST≤5.0×UNL (upper limit of normal) .

Exclusion Criteria:

Have received interventional therapy for liver cancer (except cryotherapy, radio frequency and microwave); The coagulation function is severely decreased and cannot be corrected; The main portal vein is completely embolized by cancer embolism, and the formation of collateral vessels is few; Patients with active hepatitis or severe infection who cannot be treated at the same time; Patients with cachexia or multiple organ failure;Persons with uncontrollable neurological or mental diseases or mental disorders, poor compliance, unable to cooperate and describe the treatment response; primary brain tumors or central nerve metastases have not been controlled, and have obvious intracranial hypertension or neuropsychiatric symptoms ; Pregnant or lactating women; Received other clinical trial drug treatments in the past 4 weeks; Allergy to any test drug or mannitol (excipient); Other situations where the investigator believes that the patient should not participate in this trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Estimated)
Dates: Start 2021-10 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate, ORR | 24 months
  The number of cases that achieved complete remission (CR) or partial remission (PR) accounted for the percentage of patients with evaluable efficacy.

SECONDARY OUTCOMES:
disease control rate, DCR | 24 months
  The number of complete remission (CR), partial remission (PR) and stable disease (SD) cases accounted for the percentage of patients with evaluable efficacy.
Survival rate | 24 months
  After a period of follow-up, the proportion of patients who are still alive. Observation in this study 1-year survival rate and 2-year survival rate
Time to progress, TTP | 24 months
  Time from start of TACE treatment to disease progression
Overall survival, OS | 24 months
  Time from the start of TACE treatment to death from any cause

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China